CLINICAL TRIAL: NCT04347564
Title: Usability of the Software MacuFix for the Categorization of Metamorphopsia and Evaluation of Patient Adherence Compared to the Amsler Grid
Brief Title: Usability of the Software MacuFix for the Categorization of Metamorphopsia
Acronym: MacuFix
Status: Completed | Type: Observational
Sponsor: Augenheilkunde Lindenthal (Other)
Responsible Party: Principal Investigator, Daniela Claessens, Daniela Claessens, Dr.med., M.Sc., Augenheilkunde Lindenthal
Other Study IDs: metacat; NCT04347564 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Vision Disorders
Keywords: metamorphopsia; age-related macular degeneration; diabetic macular edema; home test
MeSH Terms: conditions — Vision Disorders; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The usability of a novel test to categorize a distorted visual impression (metamorphopsia) is examined with the questionnaire "SUS"

DETAILED DESCRIPTION:
Introduction Diseases of the retinal centre (macula) can lead to a distorted visual impression (metamorphopsia). The usability of a novel on-screen test to categorize metamorphopsia is to be examined with the questionnaire "SUS" to determine how user-friendly the software is perceived.

Purpose To examine the usability of the software for persons perceiving metamorphopsia employing the questionnaire SUS.

Aim of the work Improvement of the software in terms of user-friendliness.

Methods For this observational pilot study, 30 persons are to be recruited from the patient pool of a private practice.

Primary endpoint: Score of the SUS questionnaire.

Each participating person performs the test once with each eye wearing appropriate near correction. The test shows on a screen 4 square fields with a grid pattern of horizontal and vertical lines. All 4 fields have lines that are partially distorted. The task of the test person is to select the field with more distinctively distorted lines when viewed with one eye.This selection must be made at least 10 times per eye: an algorithm determines the smallest correctly named distortion difference. Afterwards each person answers the System Usability Scale (SUS) questionnaire, SUS contains five positive and five negative statements on the usability of the system being evaluated. For each statement, the study participant gives his or her approval or rejection in the form of a scale ranging from 1= "strong approval" to 5= "strong rejection" of the statement. The results of the SUS questionnaire are used to calculate a numerical value (SUS score).

ELIGIBILITY:
Inclusion Criteria:

1. Distorted visual impression in at least one eye, detected with Amsler grid:
2. Best-corrected visual acuity (BCVA): at least 20/200; age over 18 years; presence of a declaration of consent to participate in the study

Exclusion Criteria:

No distorted visual impression in both eyes; best corrected visual acuity under 0.1; age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 persons, age at least 18 years, BVCA at least 20/200
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Claessens, MD, Principal Investigator — Augenheilkunde Lindenthal
Locations (1):
- Augenheilkunde Lindenthal, Cologne, Germany

REFERENCES:
- [Derived] Claessens D, Ichhpujani P, Singh RB. MacuFix(R) versus Amsler grid for metamorphopsia categorization for macular diseases. Int Ophthalmol. 2022 Jan;42(1):229-238. doi: 10.1007/s10792-021-02017-3. Epub 2021 Aug 22. PMID 34420124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 75 patients questioned, 45 participated in the study.
Groups:
- Initial Population: As part of a routine examination, each participating patient carried out the MacuFix test with each eye with adequate near correction once in the period 4th May, 2020 - 30th June, 2020. In addition, BCVA was measured, patients filled out the vision-related questionnaire NEI VFQ-25, patients were asked about the frequency of use of the Amsler test, a retinal examination and a spectral domain optical coherence tomography was performed. After performing the MacuFix® test all study patients filled out the questionnaire SUS. If they were interested, the patients were given a link for free use of MacuFix® as a home test or they could download the test as an app for use with an iPad or smartphone (MacuFix group). 3 months after the study day patients were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI VFQ-25 once more.
Period: Overall Study
Arm/Group | Initial Population
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Initial Population: As part of a routine examination, each participating patient carried out the MacuFix test with each eye with adequate near correction once in the period 4th May, 2020 - 30th June,2020. In addition, BCVA was measured, patients filled out the vision-related questionnaire NEI VFQ-25, patients were asked about the frequency of use of the Amsler test, a retinal examination and a spectral domain OCT was performed. After performing the MacuFix® test all study patients filled out the pseudonymised questionnaire SUS. If they were interested, the patients were given a link for free use of MacuFix® as a home test on a PC for future use of the test. Alternatively, the patients could download the test as an app for use with an iPad or smartphone. 3 months after the study day patients were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI-VFQ-25 once more.
Arm/Group | Initial Population
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants] — The mean age was 68 ± 9.7 years (SD)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 45
BCVA [Mean (Standard Deviation); unit: Snellen decimal] — best corrected visual acuity (BCVA) given as Snellen decimal
  Snellen decimal | 0.6 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Score of System Usability Scale (SUS) Questionnaire
Description: Patients filled out the SUS questionnaire immediately after completing the MacuFix test. SUS consists of ten statements each with five possible answers ranging from complete rejection to complete agreement. For each statement, the participant gives his or her approval or rejection in the form of a scale ranging from 1=strong approval to 5=strong rejection. The results of the SUS questionnaire are used to calculate a numerical value (SUS score).The results can have a value between 0 (worst application imaginable) and 100 (best application imaginable)
Time Frame: 1 day
Population: 45 patients
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Initial Population: As part of a routine examination, each participating patient carried out the MacuFix test with each eye with adequate near correction once in the period 4th May, 2020 - 30th June,2020. In addition, BCVA was measured, patients filled out the vision-related questionnaire NEI VFQ-25, patients were asked about the frequency of use of the Amsler test, a retinal examination and a spectral domain OCT was performed. After performing the MacuFix® test all study patients filled out the questionnaire SUS. If they were interested, the patients were given a link for free use of MacuFix® as a home test on a PC for future use of the test. Alternatively, the patients could download the test as an app for use with an iPad or smartphone. 3 months after the study day patients were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI-VFQ-25 once more.
Arm/Group | Initial Population
Number analyzed (Participants) | 45
score on a scale | 76.7 (15.5)

2. Secondary Outcome: Median Time Interval (in Days) Between Two Self-test Measurements (MakuFix or Amsler Respectively) to Assess the Test Adherence
Description: After a positive vote by the Ethics Committee of the North Rhine Medical Association (No. 2020057) 45 patients were included in the study from 4th May, 2020 - 30th June, 2020. Based on the amendment approval of the competent ethics committee (No. 600213225) participating persons were offered to use the App MacuFix® as a home test and to start a prospective, controlled study to examine the adherence using a self-test and evaluate the vison-related quality of life.
  On the study day and 3 months later each patient was asked about the frequency of use of the Amsler test.
  The time interval given by the patient between two Amsler Tests (Amsler group) or two MacuFix texts (MacuFix group) was assessed in days.
Time Frame: On the study day and 3 months after the study day, patients were asked how many days usually elapsed after a test with the method they chose until the next time they used this test method.
Population: difference in frequency of using the Amsler Grid or the app MacuFix® measured as the time interval (days) between two measurements to assess test adherence
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Initial Population: As part of a routine examination, each participating patient carried out the MacuFix test with each eye with adequate near correction once in the period 4th May, 2020 - 30th June,2020. In addition, BCVA was measured, patients filled out the vision-related questionnaire NEI VFQ-25, patients were asked about the frequency of use of the Amsler test, a retinal examination and a spectral domain OCT was performed. After performing the MacuFix® test all study patients filled out the questionnaire SUS. If they were interested, the patients were given a link for free use of MacuFix® as a home test on a PC for future use of the test. Alternatively, the patients could download the test as an app for use with an iPad or smartphone. 3 months after the study day patients were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI VFQ-25 once more.
Arm/Group | Initial Population
Number analyzed (Participants) | 45
days | 13 [3.82 to 23.37]

3. Secondary Outcome: Change of Vision-related Quality of Life (NEI VFQ-25, Subscale 7) After Use of the App MacuFix Versus Amsler Grid/no Test
Description: The validated questionnaire "National Eye Institute Visual Function Questionnaire-25" (NEI VFQ-25) was used to measure vision-related quality of life. The values in the questionnaire can take values from 0 to 100. High values in this questionnaire correspond to a better quality of life, low values to a poor quality of life. The 25 questions of this questionnaire can be assigned to 12 scales.
Time Frame: The validated questionnaire "National Eye Institute Visual Function Questionnaire-25" (NEI VFQ-25) was used at baseline and after 3 months.
Population: Of 45 patients included in the study, 29 subjects completed the questionnaire-25 NEI VFQ-25 before the study day and after 3 months of app use ("app user" group: 20 subjects) or 3 months of non-use ("comparison group" group: 8 performed the Amsler test, 1 did not use a self-test).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- App-users: 12-14 weeks after the study day patients using MacuFix® as a home test were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI-VFQ-25 once more.
- Amsler Grid or no Home Test: 12-14 weeks after the study day patients using the Amsler Grid as a home test or no home test were asked whether they agreed to be interviewed about the frequency of using a home test and whether they were willing to answer the questionnaire NEI-VFQ-25 once more.
Arm/Group | App-users | Amsler Grid or no Home Test
Number analyzed (Participants) | 20 | 9
score on a scale | 20.31 [10.25 to 30.37] | -3.47 [-16.24 to 9.30]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Initial Population
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
Comparability of MacuFix® and the Amsler Grid, is to some extent limited, because MacuFix® tests the central 4° of the visual field whereas the Amsler Grid examines 10° when used in the intended distance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04347564/Prot_SAP_000.pdf